CLINICAL TRIAL: NCT07111117
Title: Comparison of 18F Labeled Analog of MIBG (18F-MFBG) PET/CT and 123I-MIBG SPECT in Pediatric Patients With Neuroblastoma
Acronym: NEUROBLASTOTEP
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institut Curie (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IC 2021-11
Record Dates: First submitted 2024-01-10; First posted 2025-08-08 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-07

CONDITIONS: Neuroblastoma
Keywords: Neuroblastoma; PET / CT; Imaging; Radiotracer
MeSH Terms: conditions — Neuroblastoma

STUDY DESIGN:
Intervention Model Description: Neuroblastotep is a phase II, national, multicenter, prospective, interventional, open-label, non-randomized, single-arm pilot study (each patient being his own control). It is a concordance study comparing 18F-MFBG PET (= new diagnostic procedure) to 123I-MIBG scintigraphy (= gold standard) in neuroblastoma.
  18F-MFBG is the radiopharmaceutical product.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 18F-MFBG PET/CT imaging (Experimental): Participants will receive the 18F-MFBG tracer and undergo a PET/CT imaging.
  Interventions: Procedure: 18F-MFBG PET/CT imaging

INTERVENTIONS:
Procedure: 18F-MFBG PET/CT imaging — Participants will receive the 18F-MFBG tracer and undergo a PET/CT imaging.

SUMMARY:
The goals of the NEUROBLASTOTEP trial is to compare the diagnostics performance of a the 18F-metafluorobenzylguanidine (18F-MFBG) Positron Emission Tomography / Computed Tomography scan (PET/CT) compared to 123I-metaiodobenzylguanidine (123I-MIBG scintigraphy (current gold standard) for imaging in neuroblastoma.

DETAILED DESCRIPTION:
Neuroblastoma is one of the most common malignancies of childhood: 130 to 150 new cases are recorded each year in France. Currently, 123I-metaiodobenzylguanidine scintigraphy (123I-MIBG scan) is considered as a gold standard in neuroblastoma for assessing metastatic extension, as well as planning and evaluating response to treatment or detecting relapse. Regretfully, 123I-MIBG scintigraphy implies many disadvantages for our patients, mainly the length of the procedure (planned on two consecutive days), length of the imaging (45-90 minutes) and the required premedication for thyroid protection.

18F-metafluorobenzylguanidine (18F-MFBG) is a new specific Positron Emission Tomography (PET) tracer providing a specific Norepinephrine transporter (NET) expressing imaging with fluor-18, a routinely available radionuclide that offers higher resolution for lesion detection and shorter acquisitions for pediatric patients, and potentially lower radiation exposure.

The NEUROBLASTOTEP trial aims at demonstrating that 18F-MFBG PET/CT diagnostic performances are at least as good as 123I-MIBG scintigraphy (current gold standard imaging radiotracer in neuroblastoma).

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically proven neuroblastoma.
2. Relapsed or refractory neuroblastoma.
3. 123I-MIBG avid neuroblastoma (positive 123I-MIBG scintigraphy = showing at least one neuroblastoma lesion (either primary or metastatic) with a significant avidity for 123I-MIBG), performed within 2 weeks to 2 days prior to 18F-MFBG PET/CT.
4. No specific treatment for neuroblastoma between 123I-MIBG scintigraphy and 18F-MFBG PET/CT (PET/CT shall not delay therapeutic management.)
5. Age ≥ 365 days to < 18 years old. For children under 13 months, day of birth should be collected.
6. Weight ≥ 9 kg.
7. Performance Status: Lansky or Karnofsky ≥ 60%.
8. Signed written informed consent by the 2 holders of the parental authority or legal representative(s).
9. Patients covered by a health insurance system.

Exclusion Criteria:

1. Patient inability to comply with protocol requirements without general anesthesia.
2. Pregnant or breastfeeding patient. If indicated, at the investigator's discretion, patients of childbearing potential should have urinary pregnancy test the day of the PET/CT procedure, prior to the MFBG administration.
3. Any treatment likely to interact with MIBG initiated/modified between scintigraphy with MIBG and PET/CT with MFBG.
4. Patient with a parent or legal representative with altered mental status or psychiatric disorder that, in the opinion of the investigator, would preclude a valid informed consent

Ages: 365 Days to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2028-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Diagnostic agreement between 18F-MFBG PET/CT (new procedure) and 123I-MIBG scintigraphy (gold standard) | The day of the PET/CT procedure
  % patients in whom concordance between the 2 procedures is reached.

SECONDARY OUTCOMES:
Description of discrepancies | The day of the PET/CT procedure
  In case of non-perfect agreement, the observed discrepancies will be described. Agreement between the SIOPEN and Curie scores will be estimated.
Dosimetric comparison between the two procedures | The day of the PET/CT procedure
  One-point activity concentration measurement for normal organs (lung, liver, renal parenchyma, pancreas, spleen, adrenal gland, bladder, thyroid, heart, gonadic, eyes).
Improvement of patient management during the diagnostic procedure | The day of the PET/CT procedure
  Improvement of patient management will be evaluated by a short satisfaction survey after PET procedure, using satisfaction scales. The satisfaction and feeling variables will be described for the 123I-MIBG scintigraphy and 18F-MFBG PET/CT examinations by their repartition for the qualitative variables and by their distribution
Optimization the 18F-MFBG PET procedure (dose injected, imaging protocol) | The day of the PET/CT procedure
  PET images will be acquired in list-mode to ensure multiple reconstruction for different acquisition duration, in order to determine optimal duration.
Optimization the 18F-MFBG PET procedure (dose injected, imaging protocol) | The day of the PET/CT procedure
  PET images will be acquired in list-mode to ensure multiple reconstruction for different acquisition duration, in order to determine optimal injected activity

CONTACTS AND LOCATIONS:
Overall Officials: Tissot Hubert, MD, Principal Investigator — Institut Curie
Locations (3):
- France (3):
  - Institut Curie, Paris
  - Hôpital Armand Trousseau, Paris
  - Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: Yes
Sponsor will share de-identified data sets. Documents generated under the project will be disseminated in accordance with Institut Curie policies
Supporting Information: Study Protocol, SAP
Time Frame: Data requests can be submitted starting 9 months after last article publication and will be made accessible for up to 12 months
Access Criteria: Access to trial individual participant data can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a data sharing agreement (DSA).